CLINICAL TRIAL: NCT00609349
Title: The Early Recognition of Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-250 ex 04/05
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: risk factors for pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- connective tissue disease (Other): all patients suffer from a connective tissue disease representing a risk for the development of pulmonary hypertension
  Interventions: Device: ETED, CPET, RHC

INTERVENTIONS:
Device: ETED, CPET, RHC — exercise tricuspid echo doppler (ETED): allows the estimation of systolic pulmonary arterial pressure at exercise cardiopulmonary exercise test (CPET) allows to measures exercise capacity (peakVO2)
  right heart catheterisation (RHC): is the gold standard for the measurement of pulmonary arterial pressure values

SUMMARY:
The early detection of pulmonary arterial hypertension may help to improve prognosis of the disease. It is assumed that in the early stages of pulmonary arterial hypertension, pulmonary arterial pressure values may be normal at rest, but the remodelling of small arteries leads to stiffening resulting in increased pulmonary arterial pressure during exercise. In the present study we investigate patients with risk factors for pulmonary arterial hypertension (e.g. connective tissue disease) by combining exercise tricuspid echo doppler and cardiopulmonary exercise test to screen patients for exercise-induced pulmonary hypertension and control the results by the gold standard right heart catheterisation at rest and during exercise. We expect that using this screening method, patients with pulmonary arterial hypertension would be recognized earlier.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare, life-threatening disease. It is characterised by the elevation of pulmonary arterial pressure and pulmonary vascular resistance. A remodelling of small pulmonary vessels characterised by the proliferation of the adventitia, the hypertrophy of the media and fibrosis of the intima can be observed on the microscopic level.

According to the actual classification of Venice (2003), PAH can be idiopathic, familiar or associated to other diseases and conditions (APAH). About 15 different clinical entities belong to the APAH group: connective tissue diseases such as systemic sclerosis, mixed connective tissue disease, or systemic lupus erythematodes being among the most frequent. The development of APAH in these diseases results in decreased survival. Successful therapies include prostanoids, endothelin receptor antagonists and phosphodiesterase-5 inhibitors, however, the effects in associated conditions appear smaller compared to idiopathic PAH. The early recognition of APAH may promote better treatment results and prognosis.

Hemodynamically, PAH has been defined as a mean pulmonary arterial pressure (MPAP) > 25mmHg at rest, or > 30mmHg during exercise.

It is assumed that in the early stages of PAH, pulmonary arterial pressure values may be normal at rest, but the remodelling of small arteries leads to stiffening resulting in increased pulmonary arterial pressure during exercise (latent PAH).

Doppler echocardiography, by using the tricuspid regurgitation jet and the simplified Bernoulli-equation, is a well established clinical method for the estimation of systolic pulmonary arterial pressure at rest (rSPAP). A close correlation between rSPAP values from echo and right heart catheterisation (RHC) has been described. A promising non-invasive method to detect SPAP during exercise is Exercise Tricuspid Echo Doppler (ETED). Previous studies suggested, that SPAP during exercise can be assessed with ETED in patients with connective tissue diseases, and it was suggested that a considerable proportion of these patients suffered from latent PAH. However, the results of these studies were not controlled by the gold standard RHC. According to present guidelines, RHC is needed for the definite diagnosis of PAH, which allows the precise measurement of MPAP, pulmonary arterial wedge pressure, right atrial pressure and cardiac output, and the calculation of pulmonary vascular resistance.

Cardiopulmonary exercise testing (CPET) is a reliable method to objectively evaluate exercise capacity. Patients with latent PAH may suffer from dyspnea and early fatigue during exercise and may have a reduced exercise capacity. A low peak O2 uptake was associated with a poor prognosis in patients with PAH.

In the present study we investigate patients with risk factors for PAH by combining ETED and CPET and control the results by RHC at rest and during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis
* SLE
* Late corrected left-right shunt
* HIV Infection
* Splenectomy over 10 years
* Haemoglobinopathy and Thrombocytosis
* Ventriculo-atrial Shunt
* Liver cirrhosis/other portal Hypertension
* Anamnestic Aminorex or PhenFen abuse
* Close relatives of patients with IPAH
* Healthy controls

Exclusion Criteria:

* Known PAH
* Severe lung or bronchial disease (FEV1 <70% predicted)
* Systolic LV dysfunction (LVEF <50%) or diastolic dysfunction (pulmonary arterial "wedge" pressure (PAWP) ≥15 mmHg)
* Valvular dysfunction > Grad I (except of Tricuspidal- and Pulmonary insufficiency)
* Uncontrolled systemic arterial hypertension (rest >150 mmHg systolic or 90 mmHg diastolic; exercise >220 mmHg systolic)
* Uncontrolled ventricular arrythmia
* Uncontrolled supraventricular arrythmia
* Myocardial infarction within last 12 months
* Pulmonary embolism within last 12 months
* Significant change in therapy or larger operation within last 12 weeks
* Inability of performing exercise on cycle ergometer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
pulmonary arterial pressure | measurements with right heart catheterisation within 1 month after exercise tricuspid doppler

SECONDARY OUTCOMES:
exercise capacity (peakVO2, 6 minute walk distance) | controlled at 1 year after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria

REFERENCES:
- [Derived] Kovacs G, Maier R, Aberer E, Brodmann M, Scheidl S, Hesse C, Troester N, Salmhofer W, Stauber R, Fuerst FC, Thonhofer R, Ofner-Kopeinig P, Gruenig E, Olschewski H. Assessment of pulmonary arterial pressure during exercise in collagen vascular disease: echocardiography vs right-sided heart catheterization. Chest. 2010 Aug;138(2):270-8. doi: 10.1378/chest.09-2099. Epub 2010 Apr 23. PMID 20418368
- [Derived] Kovacs G, Maier R, Aberer E, Brodmann M, Scheidl S, Troster N, Hesse C, Salmhofer W, Graninger W, Gruenig E, Rubin LJ, Olschewski H. Borderline pulmonary arterial pressure is associated with decreased exercise capacity in scleroderma. Am J Respir Crit Care Med. 2009 Nov 1;180(9):881-6. doi: 10.1164/rccm.200904-0563OC. Epub 2009 Aug 13. PMID 19679693